CLINICAL TRIAL: NCT03265665
Title: ACTION: physicAl aCtiviTy In minOrity womeN With Asthma Intervention
Brief Title: physicAl aCtiviTy In minOrity womeN With Asthma Intervention
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sharmilee Nyenhuis, Associate Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-0466; K01HL133370 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-29 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: walking; African American women; lifestyle
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTION Intervention (Experimental): Women in the ACTION intervention will attend 1 asthma education/physical activity session and 5 group sessions in community location convenient to participants during the adoptive phase (24-weeks) and 1 group session during the maintenance phase (12-weeks). Each session will last approximately 2 hours. Participants will be given Fitbit Charge HR to monitor their daily steps and will be sent motivational, educational and reminder text messages up to 3 times per week.
  Interventions: Behavioral: ACTION Intervention
- Enhanced usual care (Other): Women in the Enhanced usual care arm will attend 1 asthma education/physical activity session and be given a Fitbit Charge HR to monitor their daily steps. They will be given a static step goal to achieve. Only reminder text messages for data collection visits will be sent.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: ACTION Intervention — The intervention is based on the Women's Lifestyle Physical Activity Program, a culturally sensitive lifestyle physical activity intervention for African American (AA) women. There are 2 phases to the intervention: Adoptive (24 weeks) and Maintenance (12 weeks). 3 motivational/reminder texts will be made each week during the adoption phase. 5 Group sessions(adoptive): Participants will be given individualized step goals, watch a short DVD featuring AA women demonstrating skills and sharing experiences of engaging in walking. 1 Group session (maintenance): watch a short DVD featuring AA women demonstrating skills and sharing experiences of engaging in walking, reinforce barriers and facilitators to walking. An interventionist will lead a discussion on role-modeling and encouraging problem solving. Each intervention group will have 10 women with 1 interventionist. Data will be collected at 3 time points: baseline, 24-weeks and 36-weeks.
  Other Names: Group sessions
  Arms: ACTION Intervention
Other: Enhanced usual care — Participants will attend 1 two hour asthma education/physical activity session at community location near them. Participants will review basic asthma topics in a didactic session and will include exercising with asthma and exercise-induced asthma. Participants will be given Fitbit and provided instructions on how to use it. Participants may receive 2 newsletters with information on asthma and reminder texts regarding data collection visits.
  Data will be collected at 3 time points: baseline, 24-weeks and 36-weeks.
  Arms: Enhanced usual care

SUMMARY:
The ACTION intervention: physicAl aCtiviTy In minOrity womeN with asthma is a 3lifestyle physical activity intervention refined to be applicable for sedentary African American (AA) women with asthma. The main outcome of this study is to test the feasibility, acceptability and estimate the efficacy of the ACTION intervention in a randomized controlled pilot of 80 AA women with asthma within a pragmatic community setting at 24-weeks.

DETAILED DESCRIPTION:
Asthma is a highly prevalent chronic disease that disproportionately impacts African American (AA) women. AA women have poorer asthma-related quality of life and higher rates of asthma exacerbations, healthcare utilization and mortality compared to Caucasian women. Further, AA women are less physically active than any other subgroup of adults, which may help explain the asthma health disparities, found between AA and Caucasian women. Physical inactivity among individuals with asthma is associated with poor asthma control and respiratory function, greater health care utilization, and poorer quality of life. Given the connection between poor asthma outcomes and physical inactivity, addressing physical activity (PA) among sedentary AA women with asthma is imperative. Physical activity demonstrated improvement in asthma outcomes specifically asthma control, quality of life and healthcare utilization. Despite these benefits, fewer than 25% of AA women with asthma engage in regular physical activity. The ACTION intervention: physicAl aCtiviTy In minOrity womeN with asthma is a lifestyle PA intervention refined to be applicable for sedentary AA women with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as female and black or AA
* Age 18-70
* Sub-optimally controlled persistent asthma based on Asthma Control Test (ACT <20)
* Wiling to enroll and provide written-informed consent
* Willing to be randomly assigned to treatment or control group

Exclusion Criteria: • Plans to relocate outside of the Chicagoland area during the study period.

* Unable to ambulate without human assistance (ie. use of a wheelchair, scooter)
* History of significant mental illness (e.g. uncontrolled bipolar disorder, psychoses)
* Currently pregnant, planning to become pregnant over the next 3 months
* Diagnosis of COPD (emphysema or chronic bronchitis) suggested by patient report of doctor diagnosis or smoking history (>20 pack years)
* Poorly controlled high blood pressure (BP >180/100 at baseline visit)
* Family/household member of another study participant or staff member
* Inability to speak, read or understand English;
* Investigator discretion for safety or protocol adherence reasons
* Participation in ACTION focus groups (Aim 1) or pre-pilot (Aim 2) of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The focus population for this study is sedentary African-American (AA) women with asthma. All participants included in the study will self-identify themselves as female and AA. This study population was chosen as AA women are disproportionately impacted by physical inactivity and asthma compared to Caucasian men and women and AA men.
Enrollment: 53 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmilee M Nyenhuis, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital and Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ACTION Intervention: Women in the ACTION intervention will attend 1 asthma education/physical activity session and 5 group sessions during the adoptive phase (24-weeks) and 1 group session during the maintenance phase (12-weeks). Each session will last approximately 2 hours. Participants will be given Fitbit Charge HR to monitor their daily steps and will be sent motivational, educational and reminder text messages up to 3 times per week.
  ACTION Intervention: The intervention is based on the Women's Lifestyle Physical Activity Program, a culturally sensitive lifestyle physical activity intervention for African American (AA) women. There are 2 phases to the intervention: Adoptive (24 weeks) and Maintenance (12 weeks). 3 motivational/reminder texts will be made each week during the adoption phase. 5 Group sessions(adoptive): Participants will be given individualized step goals, watch a short DVD featuring AA women demonstrating skills and sharing experiences of engaging in walking. 1 Group session (maintenance): watch a short DVD featuring AA women demonstrating skills and sharing experiences of engaging in walking, reinforce barriers and facilitators to walking. An interventionist will lead a discussion on role-modeling and encouraging problem solving. Each intervention group will have 10 women with 1 interventionist. Data will be collected at 3 time points: baseline, 24-weeks and 36-weeks.
- Enhanced Usual Care: Women in the Enhanced usual care arm will attend 1 asthma education/physical activity session and be given a Fitbit Charge HR to monitor their daily steps. They will be given a static step goal to achieve. Only reminder text messages for data collection visits will be sent.
  Enhanced usual care: Participants will attend 1 two hour asthma education/physical activity session. Participants will review basic asthma topics in a didactic session and will include exercising with asthma and exercise-induced asthma. Participants will be given Fitbit and provided instructions on how to use it. Participants will receive 2 newsletters with information on asthma and reminder texts regarding data collection visits.
  Data will be collected at 3 time points: baseline, 24-weeks and 36-weeks.
Period: 24-week Data Collection
Arm/Group | ACTION Intervention | Enhanced Usual Care
Started | 25 | 28
Completed | 19 | 21
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 4 | 5
Period: 36-week Data Collection
Arm/Group | ACTION Intervention | Enhanced Usual Care
Started | 23 (Used the number of participants that did not withdraw from the study. If a participant did not complete the 24 week week data collection, they were still allowed to complete the 36-week data collection. Thus the number we started with for this period was the total number of participants in each group that did not withdraw from the study.) | 26 (Used the number of participants that did not withdraw from the study. If a participant did not complete the 24 week week data collection, they were still allowed to complete the 36-week data collection. Thus the number we started with for this period was the total number of participants in each group that did not withdraw from the study.)
Completed | 17 | 18
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Usual Care: Women in the Enhanced usual care arm will attend 1 asthma education/physical activity session and be given a Fitbit Charge HR to monitor their daily steps. They will be given a static step goal to achieve. Only reminder text messages for data collection visits will be sent.
  Enhanced usual care: Participants will attend 1 two hour asthma education/physical activity session at community location near them. Participants will review basic asthma topics in a didactic session and will include exercising with asthma and exercise-induced asthma. Participants will be given Fitbit and provided instructions on how to use it. Participants may receive 2 newsletters with information on asthma and reminder texts regarding data collection visits.
  Data will be collected at 3 time points: baseline, 24-weeks and 36-weeks.
- Total: Total of all reporting groups
Arm/Group | ACTION Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.87 (11) | 43.84 (14) | 43.38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 28 | 53
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 28 | 53
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.97 (7) | 36.86 (12) | 36.44 (10)
Household Income (<$30,000/year) [Count of Participants; unit: Participants] | 17 | 15 | 32
Insurance status (medicare/medicaid/medical assistance) [Count of Participants; unit: Participants] | 17 | 20 | 37
Marital status (Single/divorced/widowed) [Count of Participants; unit: Participants] | 23 | 24 | 47
Forced Expiratory Volume in 1 second [Mean (Standard Deviation); unit: Liters] | 2.06 (0.68) | 2.04 (0.58) | 2.04 (0.63)
Forced Expiratory Volume in 1 second % predicted [Mean (Standard Deviation); unit: % predicted] | 58.64 (29) | 66.85 (24) | 62.74 (27)
Unscheduled office visits in past 6 mo (Yes) [Count of Participants; unit: Participants] | 8 | 5 | 13
Emergency Department visit(s) in the past 6 mo (yes) [Count of Participants; unit: Participants] | 5 | 7 | 12
Asthma control Questionnaire(ACQ-6) [Mean (Standard Deviation); unit: units on a scale] — Asthma control questionnaire (ACQ): The ACQ score correlates with a measure of asthma control based on the GINA/NIH criteria. ACQ includes 6 questions on symptoms, activity limitation and beta2-agonist use. Each question is scored from 0 to 6 with the total score being the average of the questions. The ACQ score ranges between 0 (well controlled) and 6 (extremely poorly controlled). Recent studies show that a score of 1.5 or more on the 7-item Asthma Control Questionnaire (ACQ) indicates that a patient has inadequate asthma control.
  units on a scale | 1.69 (0.98) | 1.83 (0.86) | 1.76 (0.91)
Asthma quality of life (AQLQ) [Mean (Standard Deviation); unit: units on a scale] — The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item questionnaire. It has 4 domains: symptoms (12 items), activity limitation (6 generic and 5 patient-specific items), emotional function (5 items), and environmental stimuli (4 items). The AQLQ items are each scored on a 7-point Likert scale, with 1 representing maximal impairment and 7 representing no impairment. Scores range 1-7, with higher scores indicating better quality of life. Total score is shown here as subdomains were not analyzed.
  units on a scale | 4.66 (1.2) | 4.6 (0.91) | 4.63 (1.03)
Daily steps [Mean (Standard Deviation); unit: steps/day] | 4737.97 (1726.55) | 4958.94 (2241.91) | 4853.98 (1991.44)
Light Physical Activity [Mean (Standard Deviation); unit: minutes/day] | 576.86 (59.92) | 272.77 (62.01) | 274.17 (70.96)
Moderate Physical Activity [Mean (Standard Deviation); unit: minutes/day] | 15.78 (18.30) | 16.67 (16.56) | 16.23 (16.74)
Vigorous Physical Activity [Mean (Standard Deviation); unit: minutes/day] | 0.63 (2.48) | 0.19 (0.76) | 0.34 (1.70)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention-Recruitment
Description: The total number of participants recruited and consented in the study.
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- Screen Participants: This is the number of participants that were screened for eligibility in the study.
Arm/Group | Screen Participants
Number analyzed (Participants) | 152
participants | 53

2. Primary Outcome: Feasibility of Intervention-Withdrawals
Description: Number of participants that withdrew from the study
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 25 | 28
Participants | 2 | 2

3. Primary Outcome: Feasibility of Lifestyle PA Intervention
Description: Number of participants that completed 24-week outcomes assessment
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 23 | 26
Participants | 19 | 21

4. Primary Outcome: Acceptability of Lifestyle PA Intervention
Description: Unabbreviated scale title: ACTION Satisfaction Scale. Acceptability was measured using a 7-point Likert scale with 1 representing not satisfied and 7 representing very satisfied. Higher scores mean more satisfied with the intervention. The range is from 1-7.
Time Frame: 24-weeks
Population: Acceptability of the intervention was measured in only intervention participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 17 | 0
units on a scale | 6.88 (0.33) |

5. Primary Outcome: Acceptability of Lifestyle PA Intervention-Qualitative Data
Description: Intervention participants were asked open-ended questions about their satisfaction with the study. Responses were written down by the participant and data collector. It is not possible to summarize the data collected from the open-ended questions in tabular form as it is qualitative data.
Time Frame: 24-weeks
Population: Intervention satisfaction was only collected in those randomized to intervention group.It is not possible to summarize the data collected from the open-ended questions in tabular form.
Arm/Group | ACTION Intervention
Number analyzed (Participants) | 0

6. Secondary Outcome: Light Physical Activity Levels
Description: as measured by accelerometer and using proprietary Actilife software
Time Frame: 24 weeks
Population: The number of participants does not equal 19 (Intervention) and 21 (EUC) as we lost a number of accelerometers in the mail or did not have adequate amount of data (A minimum of 10 hours of wear time for at least three days over a 1 week period).
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 16 | 15
minutes per day | 567.13 (79.99) | 278.66 (89.43)

7. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item questionnaire. It has 4 domains: symptoms (12 items), activity limitation (6 generic and 5 patient-specific items), emotional function (5 items), and environmental stimuli (4 items). The AQLQ items are each scored on a 7-point Likert scale, with 1 representing maximal impairment and 7 representing no impairment. Scores range 1-7, with higher scores indicating better quality of life. A total score was calculated by summing all responses for each question and then dividing by the number of items in the questionnaire (n=32). Subdomains were not reported/used.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 19 | 21
score on a scale | 5.24 (1.35) | 4.70 (1.06)

8. Secondary Outcome: Asthma Control Questionnaire (ACQ-6)
Description: Unabbreviated scale title: Asthma control questionnaire (ACQ) The ACQ score correlates with a measure of asthma control based on the GINA/NIH criteria. ACQ includes 6 questions on symptoms, activity limitation and beta2-agonist use. Each question is scored from 0 to 6 with the total score being the average of the questions. The ACQ score ranges between 0 (well controlled) and 6 (extremely poorly controlled). Recent studies show that a score of 1.5 or more on the 6-item Asthma Control Questionnaire (ACQ) indicates that a patient has inadequate asthma control.Higher scores mean poorer asthma control.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 19 | 21
score on a scale | 1.28 (1.03) | 1.87 (0.99)

9. Secondary Outcome: Daily Step Counts
Description: as measured by accelerometer
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 16 | 15
steps/day | 4372.73 (1884.90) | 5196.32 (1763.58)

10. Secondary Outcome: Moderate Physical Activity Levels
Description: as measured by accelerometer and using proprietary Actilife software
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 16 | 15
minutes per day | 16.63 (23.67) | 18.07 (13.72)

11. Secondary Outcome: Vigorous Physical Activity Levels
Description: as measured by accelerometer and using proprietary Actilife software
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | ACTION Intervention | Enhanced Usual Care
Number analyzed (Participants) | 16 | 15
minutes per day | 0.37 (1.28) | 1.14 (3.03)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | ACTION Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 2/25 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTION Intervention (N=25) | Enhanced Usual Care (N=28)
skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03265665/Prot_SAP_000.pdf